CLINICAL TRIAL: NCT01225731
Title: Randomized, Double-Blinded, Placebo-Controlled, Parallel-Design, Dose-Range Finding Study of Subcutaneous Tildrakizumab (SCH 900222/MK-3222) in Subjects With Moderate-to-Severe Chronic Plaque Psoriasis (Study P05495)
Brief Title: A Study to Determine the Optimal Dose of Tildrakizumab (SCH 900222/MK-3222) for the Treatment of Moderate-to-severe Chronic Plaque Psoriasis (P05495) (MK-3222-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05495; 2009-017272-24 (EudraCT Number); MK-3222-003 (Other: Merck Research Laboratories)
Record Dates: First submitted 2010-10-07; First posted 2010-10-21 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — tildrakizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (14):
- Part 1: Tildrakizumab 5 mg (Experimental): Participants receive tildrakizumab 5 mg, subcutaneously (SC) at Weeks 0 and 4
  Interventions: Biological: tildrakizumab
- Part 1: Tildrakizumab 25 mg (Experimental): Participants receive tildrakizumab 25 mg, SC, at Weeks 0 and 4
  Interventions: Biological: tildrakizumab
- Part 1: Tildrakizumab 100 mg (Experimental): Participants receive tildrakizumab 100 mg, SC, at Weeks 0 and 4
  Interventions: Biological: tildrakizumab
- Part 1: Tildrakizumab 200 mg (Experimental): Participants receive tildrakizumab 200 mg, SC, at Weeks 0 and 4
  Interventions: Biological: tildrakizumab
- Part 1: Placebo (Placebo Comparator): Participants receive placebo, SC, at Weeks 0 and 4
  Interventions: Drug: Placebo
- Part 2: Tildrakizumab 5 mg (Experimental): Participants receive tildrakizumab 5 mg, SC, every 12 weeks for up to 36 weeks
  Interventions: Biological: tildrakizumab
- Part 2: Tildrakizumab 25 mg (Experimental): Participants receive tildrakizumab 25 mg, SC, every 12 weeks for up to 36 weeks
  Interventions: Biological: tildrakizumab
- Part 2: Tildrakizumab 100 mg (Experimental): Participants receive tildrakizumab 100 mg, SC, every 12 weeks for up to 36 weeks
  Interventions: Biological: tildrakizumab
- Part 2: Tildrakizumab 200 mg (Experimental): Participants receive tildrakizumab 200 mg, SC, every 12 weeks for up to 36 weeks
  Interventions: Biological: tildrakizumab
- Part 3: Tildrakizumab 5 mg Follow-up (No Intervention): Participants are followed for up to 20 weeks after the last dose of study drug.
- Part 3: Tildrakizumab 25 mg Follow-up (No Intervention): Participants are followed for up to 20 weeks after the last dose of study drug.
- Part 3: Tildrakizumab 100 mg Follow-up (No Intervention): Participants are followed for up to 20 weeks after the last dose of study drug.
- Part 3: Tildrakizumab 200 mg Follow-up (No Intervention): Participants are followed for up to 20 weeks after the last dose of study drug.
- Part 3: Placebo Follow-up (No Intervention): Participants are followed for up to 20 weeks after the last dose of study drug.

INTERVENTIONS:
Biological: tildrakizumab — SC administration of tildrakizumab at assigned dose
  Other Names: SCH 900222; MK-3222
  Arms: Part 1: Tildrakizumab 100 mg; Part 1: Tildrakizumab 200 mg; Part 1: Tildrakizumab 25 mg; Part 1: Tildrakizumab 5 mg; Part 2: Tildrakizumab 100 mg; Part 2: Tildrakizumab 200 mg; Part 2: Tildrakizumab 25 mg; Part 2: Tildrakizumab 5 mg
Drug: Placebo — SC administration of Placebo
  Arms: Part 1: Placebo

SUMMARY:
This is a response-driven study of tildrakuzumab for the treatment of moderate to severe chronic plaque psoriasis. The primary study hypothesis is that one or more doses of tildrakizumab will be superior to placebo for the treatment of psoriasis.

DETAILED DESCRIPTION:
Each participant will be enrolled in the trial for approximately 72-76 weeks. Each participant will receive assigned treatment at Weeks 0 and 4 in Part I. At Week 16, the dosage of treatment the patient is assigned to may be adjusted based on the Psoriasis Area and Severity Index (PASI) 75 response (responder vs non-responder). Participants will receive study medication once every 12 weeks during Part 2 (Weeks 16 to 52); no participants will receive placebo in Part 2. Part 3 is an observational period and each subject will continue to be monitored on a monthly basis through Week 72. Subjects will not receive any study medication during Part 3.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (≥18 years of age) with a diagnosis of moderate-to-severe chronic plaque psoriasis (defined by ≥10% body surface area [BSA] involvement, "moderate" or greater score on the Physician's Global Assessment [PGA] scale, and PASI score ≥12 at Baseline)
* Participants must have a diagnosis of predominantly plaque psoriasis for ≥6 months (as determined by interview and confirmation of diagnosis through physical examination by investigator) and be considered candidates for phototherapy or systemic therapy. Participants with psoriatic arthritis may be included in the study

Exclusion Criteria:

* Nonplaque forms of psoriasis specifically erythrodermic psoriasis, predominantly pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis
* Participants who will require oral or injectable corticosteroids during the trial
* Presence of any infection requiring treatment with systemic antibiotics within 2 weeks prior to Screening, or serious infection (eg, pneumonia, cellulitis, bone or joint infections) requiring hospitalization or treatment with intravenous antibiotics within 8 weeks prior to Screening
* Participants with evidence of active or untreated latent tuberculosis (TB) according to Screening criteria specified in the protocol. (Prophylactic treatment for latent TB as per local guidelines must be initiated at least 4 weeks prior to treatment with study medication)
* Previous exposure to any agents targeting interleukin-12 (IL-12) and/or Interleukin-23 (IL-23)
* Participants with prior exposure to two or more tumor necrosis factor (TNF) antagonists with discontinuation due to lack of efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2010-10-25 (Actual); Primary Completion 2011-11-04 (Actual); Study Completion 2012-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Papp K, Thaci D, Reich K, Riedl E, Langley RG, Krueger JG, Gottlieb AB, Nakagawa H, Bowman EP, Mehta A, Li Q, Zhou Y, Shames R. Tildrakizumab (MK-3222), an anti-interleukin-23p19 monoclonal antibody, improves psoriasis in a phase IIb randomized placebo-controlled trial. Br J Dermatol. 2015 Oct;173(4):930-9. doi: 10.1111/bjd.13932. Epub 2015 Oct 15. PMID 26042589
- [Derived] Kerbusch T, Li H, Wada R, Jauslin PM, Wenning L. Exposure-response characterisation of tildrakizumab in chronic plaque psoriasis: Pooled analysis of 3 randomised controlled trials. Br J Clin Pharmacol. 2020 Sep;86(9):1795-1806. doi: 10.1111/bcp.14280. Epub 2020 Mar 25. PMID 32162721
- [Derived] Jauslin P, Kulkarni P, Li H, Vatakuti S, Hussain A, Wenning L, Kerbusch T. Population-Pharmacokinetic Modeling of Tildrakizumab (MK-3222), an Anti-Interleukin-23-p19 Monoclonal Antibody, in Healthy Volunteers and Subjects with Psoriasis. Clin Pharmacokinet. 2019 Aug;58(8):1059-1068. doi: 10.1007/s40262-019-00743-7. PMID 30915660
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05495&kw=P05495&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Part 1
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo | Part 2: Tildrakizumab 5 mg | Part 2: Tildrakizumab 25 mg | Part 2: Tildrakizumab 100 mg | Part 2: Tildrakizumab 200 mg | Part 3: Tildrakizumab 5 mg Follow-up | Part 3: Tildrakizumab 25 mg Follow-up | Part 3: Tildrakizumab 100 mg Follow-up | Part 3: Tildrakizumab 200 mg Follow-up
Started | 42 | 92 | 89 | 86 | 46 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 40 | 87 | 88 | 84 | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 5 | 1 | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not meet eligibility criteria | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo | Part 2: Tildrakizumab 5 mg | Part 2: Tildrakizumab 25 mg | Part 2: Tildrakizumab 100 mg | Part 2: Tildrakizumab 200 mg | Part 3: Tildrakizumab 5 mg Follow-up | Part 3: Tildrakizumab 25 mg Follow-up | Part 3: Tildrakizumab 100 mg Follow-up | Part 3: Tildrakizumab 200 mg Follow-up
Started | 0 (Participants could progress into Part 2) | 0 (Participants could progress into Part 2) | 0 (Participants could progress into Part 2) | 0 (Participants could progress into Part 2) | 0 (Participants could progress into Part 2; no placebo was given in Part 2) | 13 (Participants were reassigned based on PASI score at Week 16) | 94 (Participants were reassigned based on PASI score at Week 16) | 153 (Participants were reassigned based on PASI score at Week 16) | 79 (Participants were reassigned based on PASI score at Week 16) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 10 | 86 | 128 | 68 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 8 | 25 | 11 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 12 | 3 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 1 | 0 | 0 | 0 | 0
Period: Part 3
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo | Part 2: Tildrakizumab 5 mg | Part 2: Tildrakizumab 25 mg | Part 2: Tildrakizumab 100 mg | Part 2: Tildrakizumab 200 mg | Part 3: Tildrakizumab 5 mg Follow-up | Part 3: Tildrakizumab 25 mg Follow-up | Part 3: Tildrakizumab 100 mg Follow-up | Part 3: Tildrakizumab 200 mg Follow-up
Started | 0 | 0 | 0 | 0 | 0 | 0 (Participants could enter the follow-up period) | 0 (Participants could enter the follow-up period) | 0 (Participants could enter the follow-up period) | 0 (Participants could enter the follow-up period) | 10 (Not all participants entered follow-up) | 86 (Not all participants entered follow-up) | 126 (Not all participants entered follow-up) | 67 (Not all participants entered follow-up)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 80 | 116 | 60
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 10 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo | Total
Number analyzed (Participants) | 42 | 92 | 89 | 86 | 46 | 355
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (12.9) | 46.3 (13.7) | 45.5 (12.8) | 43.2 (12.6) | 45.9 (11.7) | 44.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 32 | 13 | 21 | 8 | 85
  Male | 31 | 60 | 76 | 65 | 38 | 270

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index (PASI)75 Response at Week 16
Description: The PASI score measures the severity and extent of psoriasis. Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness, and scaling of the largest psoriatic area in that region producing a Lesion Score. The percentage of the area affected by disease is then estimated, ranging from 0 = no lesions to 6 = 90-100% of the region is covered providing an Area Score. Then, the Lesion Score and Area Score for each region are multiplied, producing 4 subtotals. The 4 region subtotals are multiplied by a standardized percentage of body surface area for that region (head = 0.1, trunk = 0.3, arms=0.2, and legs = 0.4); these four region calculations are added to provide the final PASI score, ranging from 0 = no disease to 72 = maximal disease). PASI 75 response was defined as >=75% improvement in PASI score when compared to the baseline score.
Time Frame: Week 16
Population: The Full Analysis Set (FAS), all randomized participants who received >=1 dose of study drug and had a baseline and >=1 post-treatment efficacy measurement. The last non-missing post-baseline PASI score was carried forward (LOCF) unless the participant discontinued drug due to lack of efficacy, loss of response, or use of prohibited medications.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo
Number analyzed (Participants) | 42 | 90 | 89 | 86 | 45
Percentage of participants | 33.33 | 64.44 | 66.29 | 74.42 | 4.44
Statistical Analysis 1: Comparison: Part 1: Tildrakizumab 5 mg vs Part 1: Placebo; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 28.89, 95% CI 2-sided [13.41 to 44.36]
Statistical Analysis 2: Comparison: Part 1: Tildrakizumab 25 mg vs Part 1: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 60.00, 95% CI 2-sided [48.42 to 71.58]
Statistical Analysis 3: Comparison: Part 1: Tildrakizumab 100 mg vs Part 1: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 61.85, 95% CI 2-sided [50.33 to 73.37]
Statistical Analysis 4: Comparison: Part 1: Tildrakizumab 200 mg vs Part 1: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 69.97, 95% CI 2-sided [58.96 to 80.99]

2. Secondary Outcome: Percentage of Participants With a PASI 75 Response at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: The FAS, all randomized participants who received >=1 dose of study drug and had a baseline and >=1 post-treatment efficacy measurement. The last non-missing post-baseline PASI score was carried forward (LOCF) unless the participant discontinued drug due to lack of efficacy, loss of response, or use of prohibited medications.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo
Number analyzed (Participants) | 42 | 90 | 89 | 86 | 45
Percentage of participants | 23.81 | 58.89 | 60.67 | 72.09 | 4.44
Statistical Analysis 1: Comparison: Part 1: Tildrakizumab 5 mg vs Part 1: Placebo; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 19.37, 95% CI 2-sided [5.15 to 33.58]
Statistical Analysis 2: Comparison: Part 1: Tildrakizumab 25 mg vs Part 1: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 54.44, 95% CI 2-sided [42.63 to 66.26]
Statistical Analysis 3: Comparison: Part 1: Tildrakizumab 100 mg vs Part 1: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 56.23, 95% CI 2-sided [44.43 to 68.03]
Statistical Analysis 4: Comparison: Part 1: Tildrakizumab 200 mg vs Part 1: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 67.65, 95% CI 2-sided [56.42 to 78.88]

3. Secondary Outcome: Percentage of Participants With Physician's Global Assessment (PGA) of "Cleared" or "Minimal" at Week 16
Description: The PGA is used to determine the overall severity of a subject's psoriasis lesions at a given time point. Overall lesions will be graded for induration, erythema, and scaling on a scale from 0 to 5. The sum of the 3 scales will be divided by 3 to obtain the PGA score. PGA is assessed as: 0= Cleared, except for residual discoloration. 1= Minimal, majority of lesions have individual scores that average . 2 =Mild, majority of lesions have individual scores that average 2. 3= Modreate, majority of lesions have individual scores that average 3. 4= Marked, majority of lesions have individual scores that average 4. 5= Severe, majority of lesions have individual scores that average 5.
Time Frame: Week 16
Population: The Full Analysis Set (FAS), all randomized participants who received >=1 dose of study drug and had a baseline and >=1 post-treatment efficacy measurement. The last non-missing post-baseline PGA value was carried forward (LOCF) unless the participant discontinued drug due to lack of efficacy, loss of response, or use of prohibited medications.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo
Number analyzed (Participants) | 42 | 90 | 89 | 86 | 45
Percentage of participants | 33.33 | 57.78 | 61.80 | 74.42 | 2.22
Statistical Analysis 1: Comparison: Part 1: Tildrakizumab 5 mg vs Part 1: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 31.11, 95% CI 2-sided [16.22 to 46.0]
Statistical Analysis 2: Comparison: Part 1: Tildrakizumab 25 mg vs Part 1: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 55.56, 95% CI 2-sided [44.48 to 66.63]
Statistical Analysis 3: Comparison: Part 1: Tildrakizumab 100 mg vs Part 1: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 59.58, 95% CI 2-sided [48.60 to 70.55]
Statistical Analysis 4: Comparison: Part 1: Tildrakizumab 200 mg vs Part 1: Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by baseline weight (≤90 kg or >90 kg) and prior use of biologics for psoriasis (Yes/No); % Difference in Response Rate = 72.20, 95% CI 2-sided [62.02 to 82.37]

4. Secondary Outcome: Percentage of Participants With PASI 90 Response at Week 16
Description: The PASI score measures the severity and extent of psoriasis. Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness, and scaling of the largest psoriatic area in that region producing a Lesion Score. The percentage of the area affected by disease is then estimated, ranging from 0 = no lesions to 6 = 90-100% of the region is covered providing an Area Score. Then, the Lesion Score and Area Score for each region are multiplied, producing 4 subtotals. The 4 region subtotals are multiplied by a standardized percentage of body surface area for that region (head = 0.1, trunk = 0.3, arms=0.2, and legs = 0.4); these four region calculations are added to provide the final PASI score, ranging from 0 = no disease to 72 = maximal disease). PASI 90 response was defined as >=90 % improvement in PASI score when compared to the baseline score.
Time Frame: Week 16
Population: The FAS, all randomized participants who received >=1 dose of study drug and had a baseline and >=1 post-treatment efficacy measurement, and data for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo
Number analyzed (Participants) | 40 | 87 | 88 | 84 | 41
Percentage of participants | 12.50 | 25.29 | 38.64 | 52.38 | 2.44

5. Secondary Outcome: Percentage of Participants With PASI 100 Response at Week 16
Description: The PASI score measures the severity and extent of psoriasis. Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness, and scaling of the largest psoriatic area in that region producing a Lesion Score. The percentage of the area affected by disease is then estimated, ranging from 0 = no lesions to 6 = 90-100% of the region is covered providing an Area Score. Then, the Lesion Score and Area Score for each region are multiplied, producing 4 subtotals. The 4 region subtotals are multiplied by a standardized percentage of body surface area for that region (head = 0.1, trunk = 0.3, arms=0.2, and legs = 0.4); these four region calculations are added to provide the final PASI score, ranging from 0 = no disease to 72 = maximal disease). PASI 100 response was defined as 100 % improvement in PASI score when compared to the baseline score.
Time Frame: Week 16
Population: The FAS, all randomized participants who received >=1 dose of study drug and had a baseline and >=1 post-treatment efficacy measurement, and data fior this endpoint
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo
Number analyzed (Participants) | 40 | 87 | 88 | 84 | 41
Percentage of participants | 5.0 | 9.20 | 14.77 | 16.67 | 0.00

6. Secondary Outcome: PASI 75 Response Rate by Time
Description: The PASI score measures the severity and extent of psoriasis. Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness, and scaling of the largest psoriatic area in that region producing a Lesion Score. The percentage of the area affected by disease is then estimated, ranging from 0 = no lesions to 6 = 90-100% of the region is covered providing an Area Score. Then, the Lesion Score and Area Score for each region are multiplied, producing 4 subtotals. The 4 region subtotals are multiplied by a standardized percentage of body surface area for that region (head = 0.1, trunk = 0.3, arms=0.2, and legs = 0.4); these four region calculations are added to provide the final PASI score, ranging from 0 = no disease to 72 = maximal disease).PASI 75 response was defined as >=75% improvement in PASI score when compared to the baseline score at Week 2, 4, 6, 8, 12, or 16.
Time Frame: Up to 16 Weeks
Population: The FAS, all randomized participants who received >=1 dose of study drug and had a baseline and >=1 post-treatment efficacy measurement. and data for the specific Week.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo
Number analyzed (Participants) | 42 | 90 | 89 | 86 | 45
Percentage of participants
  Week 2 (n=42, 89, 89, 85, 45) | 0.00 | 1.12 | 1.12 | 0.00 | 0.00
  Week 4 (n=42, 89, 89, 85, 45) | 0.00 | 11.24 | 11.24 | 3.53 | 0.00
  Week 6 (n=40, 86, 88, 84,44) | 12.50 | 20.93 | 25.00 | 30.95 | 2.27
  Week 8 (n=40, 88, 87, 83, 43) | 12.50 | 35.23 | 47.13 | 61.45 | 4.65
  Week 12 (n=40, 87, 88, 83, 42) | 25.00 | 59.77 | 61.36 | 73.49 | 4.76
  Week 16 (n=40, 87, 88, 84, 41) | 35.00 | 65.52 | 67.05 | 76.19 | 4.88

7. Secondary Outcome: Mean Change From Baseline in PASI Score at Weeks 12 and 16
Description: The PASI score measures the severity and extent of psoriasis. Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness, and scaling of the largest psoriatic area in that region producing a Lesion Score. The percentage of the area affected by disease is then estimated, ranging from 0 = no lesions to 6 = 90-100% of the region is covered providing an Area Score. Then, the Lesion Score and Area Score for each region are multiplied, producing 4 subtotals. The 4 region subtotals are multiplied by a standardized percentage of body surface area for that region (head = 0.1, trunk = 0.3, arms=0.2, and legs = 0.4); these four region calculations are added to provide the final PASI score, ranging from 0 = no disease to 72 = maximal disease).
Time Frame: Baseline and Weeks 12 and 16
Population: The FAS, all randomized participants who received >=1 dose of study drug and had a baseline and >=1 post-treatment efficacy measurement, and data for Week 12 and Week 16.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo
Number analyzed (Participants) | 42 | 90 | 89 | 86 | 45
Score on a scale
  Week 12 | -10.2 [-12.5 to -7.9] | -14.4 [-16.0 to -12.9] | -14.1 [-15.7 to -12.5] | -14.9 [-16.5 to -13.3] | -2.2 [-4.4 to 0.00]
  Week 16 | -10.0 [-12.3 to -7.6] | -14.6 [-16.2 to -13.0] | -14.9 [-16.5 to -13.3] | -15.6 [-17.2 to -14.0] | -2.4 [-4.7 to -0.2]

8. Secondary Outcome: Percentage of Participants With PASI 50 Response at Week 16
Description: The PASI score measures the severity and extent of psoriasis. Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness, and scaling of the largest psoriatic area in that region producing a Lesion Score. The percentage of the area affected by disease is then estimated, ranging from 0 = no lesions to 6 = 90-100% of the region is covered providing an Area Score. Then, the Lesion Score and Area Score for each region are multiplied, producing 4 subtotals. The 4 region subtotals are multiplied by a standardized percentage of body surface area for that region (head = 0.1, trunk = 0.3, arms=0.2, and legs = 0.4); these four region calculations are added to provide the final PASI score, ranging from 0 = no disease to 72 = maximal disease). PASI 50 response was defined as >=50 % improvement in PASI score when compared to the baseline score.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo
Number analyzed (Participants) | 42 | 90 | 89 | 86 | 45
Percentage of participants | 57.14 | 82.22 | 82.02 | 91.86 | 8.89

9. Secondary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item questionnaire that measures how much participant skin problems have affected their life. Responses range from 0=Not at all to 3=Very much. The DLQI is broken down into 6 subscales: Symptoms and feelings (range 0-6), Daily activities (range 0-6), Leisure (range 0-6), Work and school (range 0-3), Personal relationships (range 0-6), and Treatment (range 0-3). DLQI subscales were summed to yield the DLQI total score, which could range from 0 to 30. For both DLQI subscales and DLQI total score, a higher score indicated a greater negative impact on life.
Time Frame: Week 16
Population: The FAS, all randomized participants who received >=1 dose of study drug and had a baseline and >=1 post-treatment efficacy measurement, and had data for this endpoint.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo
Number analyzed (Participants) | 40 | 87 | 88 | 83 | 42
Score on a scale | -4.9 [-7.0 to -2.8] | -9.2 [-10.6 to -7.7] | -8.5 [-9.9 to -7.1] | -8.8 [-10.3 to -7.4] | 1.0 [-1.1 to 3.0]

10. Secondary Outcome: Percentage of Participants Achieving DLQI Score of 0 or 1 at Week 16
Description: as for outcome 9
Time Frame: Week 16
Population: The FAS, all randomized participants who received >=1 dose of study drug and had a baseline and >=1 post-treatment efficacy measurement, and data for this endpoint, excluding all participants on the placebo arm.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg
Number analyzed (Participants) | 40 | 87 | 88 | 83
Percentage of participants | 32.5 | 57.47 | 52.27 | 57.83

11. Secondary Outcome: Percentage of Participants Achieving a >=5 Point Reduction in DLQI at Week 16
Description: as for outcome 9
Time Frame: Week 16
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo
Number analyzed (Participants) | 40 | 87 | 88 | 83 | 42
Percentage of participants | 52.50 | 70.11 | 64.77 | 73.49 | 19.05

12. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment.
Time Frame: Up to 72 weeks
Population: All participants receiving at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo | Part 2: Tildrakizumab 5 mg | Part 2: Tildrakizumab 25 mg | Part 2: Tildrakizumab 100 mg | Part 2: Tildrakizumab 200 mg | Part 3: Tildrakizumab 5 mg Follow-up | Part 3: Tildrakizumab 25 mg Follow-up | Part 3: Tildrakizumab 100 mg Follow-up | Part 3: Tildrakizumab 200 mg Follow-up
Number analyzed (Participants) | 42 | 91 | 89 | 86 | 45 | 13 | 94 | 153 | 79 | 10 | 86 | 126 | 67
Participants | 30 | 56 | 58 | 54 | 31 | 7 | 60 | 105 | 52 | 3 | 32 | 53 | 28

13. Primary Outcome: Number of Particpants Discontinuing Study Treatment Due to Adverse Events
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment. Participants may be discontinued from study drug due to adverse events, but remain on the study.
Time Frame: Up to 52 weeks
Population: All particpants receiving at least one dose of study drug during the treatment period.
Measure: Number; unit: Participants
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo | Part 2: Tildrakizumab 5 mg | Part 2: Tildrakizumab 25 mg | Part 2: Tildrakizumab 100 mg | Part 2: Tildrakizumab 200 mg
Number analyzed (Participants) | 42 | 91 | 89 | 86 | 45 | 13 | 94 | 153 | 79
Participants | 1 | 2 | 1 | 1 | 1 | 0 | 5 | 5 | 3

ADVERSE EVENTS:
Time Frame: Up to 72 weeks
Description: All participants who received at least one dose of tildrakizumab or placebo.
Groups:
- Placebo Follow-up: Participants who received placebo in Part 1 and did not receive additional therapy.
Arm/Group | Part 1: Tildrakizumab 5 mg | Part 1: Tildrakizumab 25 mg | Part 1: Tildrakizumab 100 mg | Part 1: Tildrakizumab 200 mg | Part 1: Placebo | Part 2: Tildrakizumab 5 mg | Part 2: Tildrakizumab 25 mg | Part 2: Tildrakizumab 100 mg | Part 2: Tildrakizumab 200 mg | Part 3: Tildrakizumab 5 mg Follow-up | Part 3: Tildrakizumab 25 mg Follow-up | Part 3: Tildrakizumab 100 mg Follow-up | Part 3: Tildrakizumab 200 mg Follow-up | Placebo Follow-up
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/91 | 1/89 | 2/86 | 0/45 | 0/13 | 5/94 | 6/153 | 3/79 | 0/12 | 1/87 | 2/137 | 2/75 | 1/2
Other Adverse Events (participants affected / at risk) | 20/42 | 35/91 | 33/89 | 30/86 | 21/45 | 7/13 | 38/94 | 64/153 | 32/79 | 3/12 | 14/87 | 29/137 | 17/75 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Tildrakizumab 5 mg (N=42) | Part 1: Tildrakizumab 25 mg (N=91) | Part 1: Tildrakizumab 100 mg (N=89) | Part 1: Tildrakizumab 200 mg (N=86) | Part 1: Placebo (N=45) | Part 2: Tildrakizumab 5 mg (N=13) | Part 2: Tildrakizumab 25 mg (N=94) | Part 2: Tildrakizumab 100 mg (N=153) | Part 2: Tildrakizumab 200 mg (N=79) | Part 3: Tildrakizumab 5 mg Follow-up (N=12) | Part 3: Tildrakizumab 25 mg Follow-up (N=87) | Part 3: Tildrakizumab 100 mg Follow-up (N=137) | Part 3: Tildrakizumab 200 mg Follow-up (N=75) | Placebo Follow-up (N=2)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonn rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Tildrakizumab 5 mg (N=42) | Part 1: Tildrakizumab 25 mg (N=91) | Part 1: Tildrakizumab 100 mg (N=89) | Part 1: Tildrakizumab 200 mg (N=86) | Part 1: Placebo (N=45) | Part 2: Tildrakizumab 5 mg (N=13) | Part 2: Tildrakizumab 25 mg (N=94) | Part 2: Tildrakizumab 100 mg (N=153) | Part 2: Tildrakizumab 200 mg (N=79) | Part 3: Tildrakizumab 5 mg Follow-up (N=12) | Part 3: Tildrakizumab 25 mg Follow-up (N=87) | Part 3: Tildrakizumab 100 mg Follow-up (N=137) | Part 3: Tildrakizumab 200 mg Follow-up (N=75) | Placebo Follow-up (N=2)
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 6 (7) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 5 (6) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute tonsilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiitis (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 3 (6) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 5 (5) | 4 (5) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (9) | 12 (14) | 13 (15) | 11 (11) | 9 (10) | 3 (4) | 24 (32) | 34 (42) | 13 (21) | 0 (0) | 6 (9) | 12 (13) | 5 (6) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (3) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (5) | 6 (7) | 4 (5) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 4 (5) | 8 (8) | 3 (3) | 1 (1) | 3 (4) | 5 (5) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 5 (8) | 6 (8) | 7 (8) | 4 (6) | 0 (0) | 3 (3) | 13 (17) | 3 (6) | 0 (0) | 1 (1) | 5 (7) | 2 (3) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 0 (0) | 4 (6) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the Sponsor. The investigator further agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication in any media that report any results of the trial. The Sponsor shall have the right to review and comment on the data analysis and presentation.